CLINICAL TRIAL: NCT03157999
Title: A Pragmatic Effectiveness-implementation Trial to Evaluate a Hospital-to-home Transitional Care Intervention Compared to Usual Care for Older Adults With Multiple Chronic Conditions and Depression
Brief Title: Community Assets Supporting Transitions (CAST)
Acronym: CAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: The Ontario Spor Support Unit (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Institute for Clinical Evaluative Sciences (Other); Laurentian University (Other); The Labarge Optimal Aging Initiative (Other)
Responsible Party: Principal Investigator, Maureen Markle-Reid, Professor and Canada Research Chair in Aging, Chronic Disease and Health Promotion Interventions, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RFHSC 2000003756
Record Dates: First submitted 2017-04-12; First posted 2017-05-17 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Comorbidity; Depressive Symptoms
Keywords: Older Adults; Transitional Care; Caregiver; Intervention
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: The proposed study design is a pragmatic randomized controlled trial (RCT). A pragmatic design applies RCT methodology in actual care settings to better inform decisions on the likely benefits, harms, and costs of real world implementation. The design is further classified as a Type II hybrid effectiveness-implementation study, which assigns equal weight to assessing program effectiveness and implementation.
Who Masked: Participant, Outcomes Assessor
Masking Description: The Research Assistant who will be collecting the outcome measures will be blinded to group allocation (intervention vs. control) for the duration of data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (CAST) (Experimental): Participants in the intervention group will receive the CAST hospital-to-home transition intervention in addition to usual care.
  Interventions: Behavioral: Intervention group (CAST)
- Control group (usual care) (No Intervention): Participants assigned to the control group will receive usual care at discharge from hospital to home.

INTERVENTIONS:
Behavioral: Intervention group (CAST) — Intervention duration is expected to be 6 months. A full-time registered nurse (RN) will function as a Care Transitions Coordinator (CTC) who works collaboratively with one local hospital and other health and non-health representatives to deliver the intervention, which includes:
  * care coordination and system navigation (including facilitating timely primary care follow-up);
  * medication management;
  * assessing the needs and risk of the participants (including in-depth assessment of depressive symptoms);
  * evidence-based management of depressive symptoms and other chronic conditions to prevent the onset and worsening of other chronic conditions;
  * patient and caregiver education; and goal setting and problem-solving therapy.
  Arms: Intervention group (CAST)

SUMMARY:
The aim of this study is to test a support program for older adults with symptoms of depression and other chronic health problems after they are discharged home from hospital. The study will be conducted in three communities in Ontario (Sudbury, Burlington, and Hamilton) and the program will be implemented with input from community members. The program will be delivered by a Registered Nurse, who will provide support to patients via home visits and telephone calls. The nurse's role will involve linking patients and their caregivers with needed services and supports, reviewing medications that the patients are taking, assessing patients' health, building the skills of patients in problem-solving and managing their care, and providing education to patients and their caregivers.

DETAILED DESCRIPTION:
Implementing transitional care interventions for older adults with depressive symptoms and multiple chronic conditions (MCC) is a pressing concern since older adults with depression face persistent health disparities. The Community Assets Supporting Transitions (CAST) research team seeks to address these health inequities, and improve health outcomes in this vulnerable and under-served population by developing and implementing an intervention that will improve patients' self-management ability, support their families and caregivers, and build capacity for primary care and other health and non-health providers to collaborate in delivering home and community services. The proposed study builds on our pilot study that evaluated a nurse-led intervention for older adult home care clients with MCC and depressive symptoms and demonstrated that the intervention was feasible and effective in reducing depressive symptoms.

The overall aim of the study is to improve care transitions in older adults with MCC and depressive symptoms. The project will address three research questions:

1. What is the effect of a new, nurse-led hospital-to-home transitional care intervention compared to usual care on health outcomes and costs for older adults with MCC and depressive symptoms?
2. How is a care transition intervention adapted and implemented in diverse settings?
3. What is required to sustain and scale up the intervention? We hypothesize that the intervention will improve health outcomes and reduce use of expensive health services compared to usual care at no additional cost, from a societal perspective.

ELIGIBILITY:
Inclusion Criteria:

* Is an adult, age 65 or older;
* Is planned for discharge from hospital to the community (this includes retirement homes and transitional care beds);
* Self-reports having a diagnosis of at least two chronic conditions;
* Is experiencing depressive symptoms, assessed using the 2-item version of the Patient Health Questionnaire (PHQ-2);
* Lives within one of the study regions (Sudbury, Burlington, or Hamilton), and is not planning to move out of the region during the trial (defined as a one-year period);
* Is capable of providing informed consent, or has a substitute decision-maker who is able to provide informed consent on his/her behalf; and
* Is competent in English, or has an interpreter who is competent in English.

Exclusion Criteria:

* Is being discharged from the hospital to a long-term care home or tertiary care.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 127 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Change in mental functioning of the older adult study participant | T1 = Baseline data collection; T2 = 6 months after randomization; T3 = 12 months after randomization
  Measured by the mental component summary (MCS) score of the Veterans RAND 12 item Health Survey (VR-12).

SECONDARY OUTCOMES:
Change in mental functioning of the family/friend caregiver of older adult participant (if applicable). | T1 = Baseline data collection; T2 = 6 months after randomization; T3 = 12 months after randomization
  Measured by the mental component summary (MCS) score of the Veterans RAND 12 item Health Survey (VR-12).
Change in physical function of the: 1) older adult study participant, 2) family/friend caregiver of older adult participant (if applicable). | T1 = Baseline data collection; T2 = 6 months after randomization; T3 = 12 months after randomization
  Measured by the physical component summary (PCS) score of the Veterans RAND 12 item Health Survey (VR-12).
Change in health-related quality of life of the: 1) older adult study participant, 2) family/friend caregiver of older adult participant (if applicable). | T1 = Baseline data collection; T2 = 6 months after randomization; T3 = 12 months after randomization
  Measured by the Veterans RAND 12 item Health Survey (VR-12).
Change in depressive symptoms of the: 1) older adult study participant, 2) family/friend caregiver of older adult participant (if applicable). | T1 = Baseline data collection; T2 = 6 months after randomization; T3 = 12 months after randomization
  As measured by the CESD-10 to determine the presence and severity of depressive symptoms.
Change in anxiety of the: 1) older adult study participant, 2) family/friend caregiver of older adult participant (if applicable). | T1 = Baseline data collection; T2 = 6 months after randomization; T3 = 12 months after randomization
  As measured by the GAD-7 (24).
Change in caregiver strain of the family/friend caregiver of the older adult study participant (if applicable) | T1 = Baseline data collection; TT2 = 6 months after randomization; T3 = 12 months after randomization
  As measured by the Modified Caregiver Strain Index
Change in utilization of health and social services by the: 1) older adult study participant, 2) family/friend caregiver of the older adult study participant. | T1 = Baseline data collection; T2 = 6 months after randomization; T3 = 12 months after randomization
  As measured by the Health and Social Services Utilization Inventory
Change in utilization of health services by the older adult study participant | T2 = 6 months after randomization; T3 = 12 months after randomization
  As identified through Institute for Clinical Evaluative Sciences (ICES) databases
Change in unmet care needs of the: 1) older adult study participant, 2) family/friend caregiver of older adult participant (if applicable). | T1 = Baseline data collection; T2 = 6 months after randomization
  As measured through the Unmet Care Needs questionnaire (developed using input from patient/caregiver co-researchers to ensure the inclusion of outcomes that are relevant and meaningful to patients and caregivers).
Change in patient-provider communication of the: 1) older adult study participant, 2) family/friend caregiver of older adult participant (if applicable). | T1 = Baseline data collection; T2 = 6 months after randomization
  As measured through the Patient-Provider Communication (PCC) questionnaire.
Change in patient-reported experience (CCCQ) for the: 1) older adult study participant, 2) family/friend caregiver of older adult participant (if applicable). | T1 = Baseline data collection; T2 = 6 months after randomization
  As measured through the adapted Client-Centred Care Questionnaired (CCCQ).
Change in patient-reported experience (IC-PREMs) for the: 1) older adult study participant, 2) family/friend caregiver of older adult participant (if applicable). | T1 = Baseline data collection; T2 = 6 months after randomization
  As measured through the adapted Integrated Care Patient-Reported Experience Measures (IC-PREMs).

CONTACTS AND LOCATIONS:
Overall Officials: Maureen F Markle-Reid, Ph.D., Principal Investigator — McMaster University; Carrie McAiney, Ph.D., Principal Investigator — University of Waterloo
Locations (4):
- Canada (4):
  - Joseph Brant Hospital, Burlington, Ontario
  - Health Sciences North/Laurentian University, Greater Sudbury, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - School of Nursing, McMaster University, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Markle-Reid M, McAiney C, Forbes D, Thabane L, Gibson M, Browne G, Hoch JS, Peirce T, Busing B. An interprofessional nurse-led mental health promotion intervention for older home care clients with depressive symptoms. BMC Geriatr. 2014 May 10;14:62. doi: 10.1186/1471-2318-14-62. PMID 24886344
- [Background] Markle-Reid MF, McAiney C, Forbes D, Thabane L, Gibson M, Hoch JS, Browne G, Peirce T, Busing B. Reducing depression in older home care clients: design of a prospective study of a nurse-led interprofessional mental health promotion intervention. BMC Geriatr. 2011 Aug 25;11:50. doi: 10.1186/1471-2318-11-50. PMID 21867539
- [Derived] Markle-Reid M, McAiney C, Fisher K, Ganann R, Gauthier AP, Heald-Taylor G, McElhaney JE, McMillan F, Petrie P, Ploeg J, Urajnik DJ, Whitmore C. Effectiveness of a nurse-led hospital-to-home transitional care intervention for older adults with multimorbidity and depressive symptoms: A pragmatic randomized controlled trial. PLoS One. 2021 Jul 26;16(7):e0254573. doi: 10.1371/journal.pone.0254573. eCollection 2021. PMID 34310640
- [Derived] Markle-Reid M, McAiney C, Ganann R, Fisher K, Gafni A, Gauthier AP, Heald-Taylor G, McElhaney J, Ploeg J, Urajnik DJ, Valaitis R, Whitmore C. Study protocol for a hospital-to-home transitional care intervention for older adults with multiple chronic conditions and depressive symptoms: a pragmatic effectiveness-implementation trial. BMC Geriatr. 2020 Jul 10;20(1):240. doi: 10.1186/s12877-020-01638-0. PMID 32650732
- See also: Ontario SPOR support unit — http://ossu.ca/